CLINICAL TRIAL: NCT02082652
Title: A Pharmacokinetic Evaluation of Etonogestrel (ENG) Implant and Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)-Based Antiretroviral Therapy in HIV-Infected Ugandan Women
Brief Title: A Pharmacokinetic Evaluation of Etonogestrel (ENG) Implant and Antiretroviral Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Catherine Chappell, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO14010195
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: HIV; Contraception
Keywords: Etonogestrel; Efavirenz; Nevirapine; Pharmacokinetics
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No ART) (Active Comparator): Etonogestrel implant in participants not yet receiving ART (control group)
  Interventions: Drug: Etonogestrel
- Nevirapine-based ART group (Active Comparator): Etonogestrel implant in participants receiving nevirapine (NVP)-based ART
  Interventions: Drug: Etonogestrel
- Efavirenz-based ART group (Active Comparator): Etonogestrel implant in participants receiving efavirenz (EFV)-based ART
  Interventions: Drug: Etonogestrel

INTERVENTIONS:
Drug: Etonogestrel — Etonogestrel single-rod subdermal implant (68mg/rod) is placed upon enrollment (day 0) and remains in place until participant requests removal or for the duration of active drug (currently approved for 3 years of use).
  Other Names: Implanon; Nexplanon

SUMMARY:
Antiretroviral therapy (medicines used to treat HIV) can interact with hormonal contraceptives which might decrease their effectiveness. The single-rod etonogestrel contraceptive implant is being more commonly used in low- and middle-income countries because if the ease of insertion and removal. Efavirenz and nevirapine are first-line HIV medicines in Sub-Saharan Africa and this study will help determine an effective way to use these medicines with the etonogestrel implant. The investigators hypothesize that women receiving nevirapine- or efavirenz-based antiretroviral therapy will have lower etonogestrel levels in their blood after six months of insertion as compared to women not taking antiretroviral therapy.

DETAILED DESCRIPTION:
Modern contraceptive use by HIV-infected women not only prevents pregnancy-related complications and economic disparity, but also prevents perinatal HIV transmission. Despite the clear benefits of highly effective modern contraceptives, there are significant unanswered questions about their safety in women infected with HIV, particularly women who are on anti-retroviral therapy (ART). Currently, non-nucleoside reverse transcriptase inhibitors (NNRTIs), such as nevirapine (NVP) and efavirenz (EFV), are the most widely prescribed HIV medications in sub-Saharan Africa and recently the WHO recommended the EFV-based ART be recommended as first-line therapy for HIV-1 infected adults, including women of reproductive age. Contraceptive implants are becoming increasingly available and popular in sub-Saharan Africa, and the etonogestrel (ENG) implant is a single rod, making insertion and removal easier than other contraceptive implants. The clinical data on concurrent use of NNRTIs and the ENG implant are limited to six case reports of contraceptive failures in the setting of EFV-based ART, highlighting the potential for a clinically significant drug-drug interaction. The investigators aim to perform a pharmacokinetic (PK) study evaluating the interaction between the ENG implant and NNRTI-based ART. The investigators propose a non-randomized, open-label, parallel, three-group, sparse-sampling PK study to compare ENG PK parameters between a control group (no ART) and two treatment groups (EFV- or NVP-based ART) in 60 HIV-1 infected women, 20 women in each group. The primary endpoint is the comparison of the mean ENG concentrations at month 6 between the control group and NNRTI treatment groups. The investigators hypothesize that women in the EFV-based and NVP-based ART group will have a significantly lower mean ENG concentration 6 months post-implant insertion, as compared to women in the control group. The investigators also aim to: 1) predict the disposition of ENG in women on NNRTI-based ART over the subsequent 2.5 years of intended use through PK modeling of ENG concentrations beyond 6 months of use in HIV-infected women, 2) estimate the long-term impact of chronic ENG exposure on EFV or NVP concentrations measured before and during 6 months of combined use, and 3) compare side-effect frequencies of the ENG subdermal implant in women not on ART and on concomitant NNRTI-based ART. The results will guide clinicians caring for HIV-infected women on whether using NNRTI-based therapy together with the ENG implant will jeopardize contraceptive efficacy due to a reduction in ENG exposure.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study
* Display willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Age between 18 and 45 years and female sex
* Diagnosis of HIV-1 infection
* Desiring ENG subdermal implant as a contraceptive method
* Participants not yet eligible for ART (based on the Ugandan Treatment Guidelines); or participants receiving NVP or EFV-based ART for a minimum of 1 month prior to screening
* Participants on EFV-based ART must have an alternative form on effective non-hormonal contraception, such as surgical sterilization or copper intrauterine device in place

Exclusion Criteria:

* For potential participants on ART: HIV-1 RNA > 400 copies/mL at screening visit
* Serum hemoglobin < 9.0 g/dl
* Elevations in serum levels of alanine transaminase (ALT) above 5 times the upper limit of normal
* Elevations in serum creatinine above 2.5 times the upper limit of normal
* Use of drugs known to be contraindicated with ENG, NVP (for women taking NVP-based ART), or EFV (for women taking EFV-based ART) within 30 days of study entry. Due to the dynamic nature of drug interactions related to antiretroviral therapy, the study team will review all concomitant medications at screening based on the US Department of Health and Human Services drug interaction table.
* Currently pregnant or postpartum <30 days at study entry. Participants must have a negative urine pregnancy test and report no unprotected sex since the last menstrual period or in the last two weeks.
* Concurrent use of other hormonal contraception (Note: use of other forms of hormonal contraception is permissible until time of study enrollment/insertion of ENG implant. Transition from other forms of hormonal contraception to ENG subdermal implant will be accommodated according to ENG product labeling.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Etonogestrel plasma concentrations | 6 months after the implant is placed

SECONDARY OUTCOMES:
NNRTI plasma concentrations | Over 6 months (baseline, Month 1, 3, and 6)
  Applies only to participants being treated with either efavirenz- or nevirapine-based antiretroviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Chappell, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chappell CA, Lamorde M, Nakalema S, Chen BA, Mackline H, Riddler SA, Cohn SE, Darin KM, Achilles SL, Scarsi KK. Efavirenz decreases etonogestrel exposure: a pharmacokinetic evaluation of implantable contraception with antiretroviral therapy. AIDS. 2017 Sep 10;31(14):1965-1972. doi: 10.1097/QAD.0000000000001591. PMID 28692531
- [Derived] Neary M, Chappell CA, Scarsi KK, Nakalema S, Matovu J, Achilles SL, Chen BA, Siccardi M, Owen A, Lamorde M. Effect of patient genetics on etonogestrel pharmacokinetics when combined with efavirenz or nevirapine ART. J Antimicrob Chemother. 2019 Oct 1;74(10):3003-3010. doi: 10.1093/jac/dkz298. PMID 31299074